CLINICAL TRIAL: NCT05286008
Title: Impact of Ultrasound-Guided Transversus Abdominis Plane Block on Postoperative Nausea and Vomiting and Early Outcome After Laparoscopic Bariatric Surgery: a Randomized Double-Blinded Controlled Trial
Brief Title: Effect of Ultrasound-guided Transversus Abdominis Plane Block After Laparoscopic Bariatric Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Guolin Wang, Professor, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GWang022
Record Dates: First submitted 2022-01-24; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Postoperative Nausea and Vomiting; Postoperative Pain
Keywords: Ropivacaine; Transversus abdominis plane block; opioid consumption; Dexamethasone
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Pain, Postoperative | interventions — Saline Solution; Sodium Chloride; Ropivacaine; Dexamethasone

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double (Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal Saline (Placebo Comparator): Before the induction of anesthesia, normal saline is used for bilateral transversus abdominis plane block in a volume of 20 mL of each side.
  Interventions: Drug: Normal saline
- Ropivacaine at high concentration (Experimental): Before the induction of anesthesia, 0.375% Ropivacaine is used for bilateral transversus abdominis plane block in a volume of 20 mL of each side
  Interventions: Drug: Ropivacaine at high concentration
- Ropivacaine and dexamethasone (Experimental): Before the induction of anesthesia, 0.375% Ropivacaine and 5.0mg dexamethasone are used for bilateral transversus abdominis plane block in a volume of 20 mL of each side
  Interventions: Drug: Ropivacaine and dexamethasone

INTERVENTIONS:
Drug: Normal saline — Before the induction of anesthesia, normal saline is used for bilateral transversus abdominis plane block in a volume of 20 mL of each side
  Other Names: 0. 9% Sodium Chloride Injection
  Arms: Normal Saline
Drug: Ropivacaine at high concentration — Before the induction of anesthesia,0.375% ropivacaine is used for bilateral transversus abdominis plane block in a volume of 20 mL of each side
  Other Names: Ropivacaine Hydrochloride Injection
  Arms: Ropivacaine at high concentration
Drug: Ropivacaine and dexamethasone — Before the induction of anesthesia, 0.375% Ropivacaine and 5.0mg dexamethasone are used for bilateral transversus abdominis plane block in a volume of 20 mL of each side
  Other Names: Ropivacaine Hydrochloride Injection
  Arms: Ropivacaine and dexamethasone

SUMMARY:
To explore and compare Ultrasound-Guided Transversus Abdominis Plane Block on Postoperative nausea and vomiting and Early Outcome After Laparoscopic Bariatric Surgery To evaluate and examine TAPB can reduce the application of intraoperative and postoperative opioids and the duration of analgesia

DETAILED DESCRIPTION:
Poor postoperative nausea and vomiting control is a leading factor that hinders the physical rehabilitation, and causes acute cognitive impairment and chronic pain syndrome. Recently, the multimodal analgesia strategies to minimise opioid-related side effects are highly desirable in open surgical procedures. The transversus abdominis plane block is a novel technique involving injection of local anaesthetic between the internal oblique and the transversus abdominis muscles of the abdominal wall. Although ropivacaine is most commonly used for this technique, the analgesic duration remains not dissatisfied. Herein, investigators will evaluate the efficacy of ultrasound-guided transversus abdominis plane(USG- TAP) block with ropivacaine in Laparoscopic Bariatric Surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is scheduled to undergo Laparoscopic Bariatric Surgery
2. Subject's American Society of Anesthesiologists physical status is I-III.
3. BMI>35kg/m2
4. The subject's parent/legally authorized guardian has given written informed consent to participate

Exclusion Criteria:

1. Subject has a diagnosis of renal or liver failure.
2. Subject has a diagnosis of mental illness
3. Subject is allergy and contraindication to Ropivacaine.
4. Subject has a history of chronic pain, a history of alcohol or opioid abuse, pre-existing therapy with opioids, intake of any analgesic drug within 48 hours before surgery.
5. Subject has any contraindication for the use
6. Subject is pregnant or breast-feeding.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-03-18 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-10-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative nausea and vomiting | 72 hours after surgery
  The Apfel score was recorded for evaluating risk for developing postoperative nausea and vomiting (PONV).

SECONDARY OUTCOMES:
cumulative Sufentanyl Consumption during surgery | during surgery
  Each patient was administered sufentanil for analgesic during surgery
cumulative Sufentanyl Consumption after surgery | 48 hours after surgery
  Each patient was administered analgesics using a PCA pump containing sufentanil (100μg) in normal saline at a totalvolume of 100 ml after leaving PACU. This device was set to deliver a basal infusion of 2 ml/h and bolus doses of 0.5ml with a 15-min lockout period. Sufentanyl cumulative consumption is recorded 24 hours postoperative
Time of First Postoperative Analgesic Requiremen | 1hour after surgery
  First postoperative pain (NRS≥5) is initially controlled by titration of sufentany
Total Dose of First Postoperative Analgesic Requirement | 1hour after surgery
  First postoperative pain (NRS≥5) is initially controlled by titration of sufentanyl.
The incidence of Side Effects | 48 hours after surgery
  The number of patients with side effects including nausea, vomiting, dizziness, headache, shivering, and pruritus is recorded for 48 hours postoperatively
Apfel score | The 1 day before the surgery
  The Apfel score was recorded for evaluating risk for developing postoperative nausea and vomiting (PONV).
Time to ambulation | 12 hours after surgery
  The obesity's time to ambulation after surge
Mean time until passage of flatus | 72 hours after surgery
  Gastrointestinal motility was evaluated by recording mean time until passage of flatus
Diffusion area of local anesthetics after transversus abdominis plane block | 30 minutes after transversus abdominis plane block
  Diffusion area of local anesthetics after transversus abdominis plane block was calculated under ultrasound assistance.
Normalized Area of Hyperalgesia Around the Incision | 48 hours after surgery
  The skin around the incision is stimulated in steps of 5 mm at intervals of 1 s starting outside of the hyperalgesic area in the direction of the incision. The distance from the incision to the first point where a 'painful', 'sore' or 'sharper'feeling occurred is measured and noted. This measurement is repeated at predefined radial lines around the incision. To eliminate the variable length of incision, this length is subtracted from the longer diameter leaving four radial distances from the end and from the middle of the incision. The normalized area of hyperalgesia is calculated by summing up the areas of the remaining four triangles measured by and Von Frey filament.

CONTACTS AND LOCATIONS:
Overall Officials: Guolin Wang, MD, Study Director — Tianjin Medical University General Hospital

IPD SHARING:
Plan to Share IPD: No